CLINICAL TRIAL: NCT06763354
Title: An Exploratory Clinical Study of the Efficacy of Gallium[68Ga]NOTA-DNA Multivalent SGC8 Injection for Bladder Tumour Imaging
Brief Title: The Efficacy of Gallium[68Ga]NOTA-DNA Multivalent SGC8 Injection for Bladder Tumour Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liu Peifeng, Principal Investigator, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIT-2024-0231
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Combination Product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with bladder tumors (Experimental)
  Interventions: Radiation: Gallium[68Ga]NOTA-DNA Multivalent SGC8 Injection

INTERVENTIONS:
Radiation: Gallium[68Ga]NOTA-DNA Multivalent SGC8 Injection — On the examination bed, the patient was placed in the lying truncated position, the perineum was disinfected with a towel, and a double-lumen urinary catheter was inserted via the perineum.Inject 50ml saline to clean the bladder once, open the drainage bag to drain.1mci SGC8 was dissolved in 50ml physiological saline. The drainage bag was clamped shut and 50ml of developer was injected into the bladder through the catheter, followed by 10ml of gas or saline (all developer in the ureter was injected into the bladder. The catheter was closed for 1 hour, during which time the patient was placed in the flat position, left lateral position, right lateral position, and supine position changing positions every 15 minutes.After 1 hour, the drainage bag was opened, the bladder was emptied with radioactive fluid, and the urine bag was replaced.

SUMMARY:
The study was planned to include patients with bladder tumors attending the Department of Urology, Renji Hospital, Shanghai Jiaotong University School of Medicine, from 09/2024 to 12/2025. Patient demographics will be collected, patients will be monitored for medical history and co-morbidities, co-morbid medications or treatments, vital signs, and cystoscopy will be performed. Patients meeting the inclusion criteria will be included in this study. Patients will receive PET/MR imaging after bladder instillation of [68Ga] NOTA-DNA multivalent SGC8 injection to assess the effectiveness of bladder tumor imaging and to evaluate the safety of [68Ga] NOTA-DNA multivalent SGC8.

The primary study was the ability of gallium [68Ga] NOTA-DNA multivalent SGC8 injection to provide tumor-specific imaging of bladder tumor patients of different genders, with a compliance rate of more than 80% when compared to the gold standard TUR pathology. To study the safety of gallium[68Ga] NOTA-DNA multivalent SGC8 injection; to assess the correlation between gallium[68Ga] NOTA-DNA multivalent SGC8 imaging ability and clinical parameters; to study the ability of gallium [68Ga]NOTA-DNA multivalent SGC8 to differentiate between bladder tumor foci and inflammatory foci; to explore the gallium [68Ga]NOTA- DNA multivalent SGC8 target PTK7 receptor protein expression in bladder tumors and the correlation between tumor differentiation and malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary enrolment with signed informed consent
2. Age >18 years, <85 years
3. Cystoscopic diagnosis of bladder tumour with imaging and pathology reports not required
4. Willingness and ability to follow trial protocol requirements.

Exclusion Criteria:

1. Pregnancy, breastfeeding, severe hepatic, renal insufficiency and children
2. Hypersensitivity to the test drug, allergy or allergy to multiple drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor specific lighting ability of Gallium[68Ga]NOTA-DNA Multivalent SGC8 | 2 year
  Number of patients whose tumors are lightened under PET/MR with Gallium[68Ga]NOTA-DNA Multivalent SGC8

SECONDARY OUTCOMES:
Safety of Gallium[68Ga]NOTA-DNA Multivalent SGC8 | 2 Year
  Adverse events within 24 hours of intravesical irrigation; Serious adverse events within 5 days of intravesical irrigation
Accuracy in clinical parameters of Gallium[68Ga] NOTA-DNA multivalent SGC8 | 2 Year
  Correlation between gallium[68Ga] NOTA-DNA multivalent SGC8 images and clinical parameters
Foci-distinguishing ability of Gallium [68Ga]NOTA-DNA multivalent SGC8 | 2 Year
  The ability of gallium [68Ga]NOTA-DNA multivalent SGC8 to differentiate between bladder tumor foci and inflammatory foci
The expression of PTK7 in bladder tumor tissues | 2 Year
  The expression of [68Ga]-NOTA-SGC8 target PTK7 receptor protein in bladder tumor tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided